CLINICAL TRIAL: NCT04637841
Title: Comparasion of the Immediate Effect of Myofascial Relaxation Technique and Kinesiology Taping on Biomechanical and Viscoelastic Properties of Plantar Fascia and Plantar Pressure Distribution in Diabetes Patients
Brief Title: Comparasion of the Immediate Effect of Myofascial Relaxation Technique and Kinesiology Taping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09.2020.948
Record Dates: First submitted 2020-11-08; First posted 2020-11-20 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus; Plantar Fascia
Keywords: stiffness; creep; plantar fascia; diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Diabetes Mellitus Kinesiology Taping Group (Active Comparator): Kinesiology tape will be applied to the left foot of the participants in diabetes mellitus group.
  Interventions: Other: Kinesiology Taping Appliying
- Kinesiology Taping Control Group (Active Comparator): Kinesiology tape will be applied to the left foot of the healthy participants in the control group.
  Interventions: Other: Kinesiology Taping Appliying
- Diabetes Mellitus Myofascial Release Group (Active Comparator): Myofascial Release Technique will be applied to the right foot of the participants in diabetes mellitus group.
  Interventions: Other: Myofascial Release Technique Appliying
- Myofascial Release Control Group (Active Comparator): Myofascial Release Technique taping will be applied to the right foot of the healthy participants in the control group.
  Interventions: Other: Myofascial Release Technique Appliying

INTERVENTIONS:
Other: Kinesiology Taping Appliying — Kinesiology tape will be applied to left foot plantar fascia of the participants in diabetes mellitus and control group.
  During taping, participants will lie in the prone position while the knee joint will be kept 90 degrees of flexion and the ankle joint in a neutral position. A "Palm Shape" taping procedure will be applied to the plantar fascia.
  Arms: Diabetes Mellitus Kinesiology Taping Group; Kinesiology Taping Control Group
Other: Myofascial Release Technique Appliying — Myofascial release technique will be applied (during 5 minutes) to right foot plantar fascia of the participants in diabetes mellitus and control group
  During appliying technique, participants will lie in the prone position while the knee joint will be kept 90 degrees of flexion and the ankle joint in a neutral position.
  Arms: Diabetes Mellitus Myofascial Release Group; Myofascial Release Control Group

SUMMARY:
As a result of glycation of collagen fibers in diabetes mellitus, an increase in thickness and stiffness is observed in the plantar fascia, which is a connective tissue. These changes in the plantar fascia affect the windlass mechanism of the foot, normal range of motion and foot plantar pressure distribution. These biomechanical effects may cause the development of diabetic foot ulcers in the later stages of the disease. We hypothesis that myofascial release technique and kinesiology taping methods have an effect on plantar fascia stiffness and plantar pressure distribution in diabetic patients. The aim of this study is to investigate the immediate effects of the two methods on the stiffness of the plantar fascia and foot sole pressure distribution in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Those with diabetic foot ulcer development risk groups 1 and 2 according to the International Working Group on the Diabetic Foot (IWGDF)
* Those who have diabetes for at least 5 years
* Ambulation independently without using an assistive device

Exclusion Criteria:

* Those with foot posture deformity
* Having another disease that will affect connective tissue properties
* Presence of orthopedic or neurological disorders that will affect plantar load distribution
* History of surgery and fractures from the ankle-foot in the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
Evaluation of foot plantar pressure distribution | Change from baseline plantar presure distrubution at following kinesiologic tape appliying and at 30min.
  Plantar pressure distrubution (gr/ cm²) on the force platform will be measured.
Evaluation of stiffness | Change from baseline stiffness of the plantar fascia at following kinesiologic tape appliying and at 30min.
  Stiffness (N/m) of the plantar fascia will be mesured using a digital handheld myometer (MyotonPro, Myoton AS, Tallinn, Estonia).
Evaluation of decrement | Change from baseline decrement properties of the plantar fascia at following kinesiologic tape appliying and at 30min.
  Decrement of the plantar fascia will be mesured using a digital handheld myometer (MyotonPro, Myoton AS, Tallinn, Estonia).
Evaluation of creep | Change from baseline creep properties of the plantar fascia at following kinesiologic tape appliying and at 30min.
  Creep of the plantar fascia will be mesured using a digital handheld myometer (MyotonPro, Myoton AS, Tallinn, Estonia).
Evaluation of relaxation time | Change from baseline relaxation time properties of the plantar fascia at following kinesiologic tape appliying and at 30min.
  Relaxation time of the plantar fascia will be mesured using a digital handheld myometer (MyotonPro, Myoton AS, Tallinn, Estonia).

SECONDARY OUTCOMES:
Evaluation of range of motion of ankle | Change from baseline range of motion at following kinesiologic tape appliying and at 30min.
  Range of motion of ankle was measured with goniometer
Evaluation of foot sole pain | Change from baseline foot sole pain at following kinesiologic tape appliying and at 30min.
  Pain was evaluated by Visual Analog Scale between 0 (no pain) and 10 (the most severe pain).
Evaluation of skin temperature | Change from baseline foot sole temperature at following kinesiologic tape appliying and at 30min.
  Plantar skin temperature will be measured by thermal imaging machine (Flir Sistem, ThermaCAM, Sweden)

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - İstanbul Medeniyet City, Istanbul
  - İstanbul Medeniyet University, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ajimsha MS, Binsu D, Chithra S. Effectiveness of myofascial release in the management of plantar heel pain: a randomized controlled trial. Foot (Edinb). 2014 Jun;24(2):66-71. doi: 10.1016/j.foot.2014.03.005. Epub 2014 Mar 21. PMID 24703512
- [Result] American Diabetes Association. 16. Diabetes Advocacy: Standards of Medical Care in Diabetes-2019. Diabetes Care. 2019 Jan;42(Suppl 1):S182-S183. doi: 10.2337/dc19-S016. PMID 30559242
- [Result] Bernard V, Staffa E, Mornstein V, Bourek A. Infrared camera assessment of skin surface temperature--effect of emissivity. Phys Med. 2013 Nov;29(6):583-91. doi: 10.1016/j.ejmp.2012.09.003. Epub 2012 Oct 18. PMID 23084004
- [Result] Chen TL, Wong DW, Peng Y, Zhang M. Prediction on the plantar fascia strain offload upon Fascia taping and Low-Dye taping during running. J Orthop Translat. 2019 Aug 7;20:113-121. doi: 10.1016/j.jot.2019.06.006. eCollection 2020 Jan. PMID 31908942
- [Result] Hicks CL, von Baeyer CL, Spafford PA, van Korlaar I, Goodenough B. The Faces Pain Scale-Revised: toward a common metric in pediatric pain measurement. Pain. 2001 Aug;93(2):173-183. doi: 10.1016/S0304-3959(01)00314-1. PMID 11427329
- [Result] Kong PW, Chua YH, Kawabata M, Burns SF, Cai C. Effect of Post-Exercise Massage on Passive Muscle Stiffness Measured Using Myotonometry - A Double-Blind Study. J Sports Sci Med. 2018 Nov 20;17(4):599-606. eCollection 2018 Dec. PMID 30479528